CLINICAL TRIAL: NCT06270407
Title: The Effect of Topical Tranexamic Acid on Postoperative Complications in Soft Tissue Plastic Surgery - A Multicenter Randomized Controlled Trial
Brief Title: The Effect of Local Application of Tranexamic Acid Versus Placebo on Postoperative Complications in Plastic Surgery
Acronym: TRANOP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Smerud Medical Research International AS (Other); Sykehuset Asker og Baerum (Other); Oslo University Hospital (Other); Sykehuset Telemark (Other Government); Sykehuset Innlandet HF (Other); Molde Hospital (Other); Haukeland University Hospital (Other); Haraldsplass Deaconess Hospital (Other); Helse Stavanger HF (Other Government); University Hospital of North Norway (Other); Bodø sykehus (Unknown); Helsinki University Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 270777; 2022-001580-28 (EudraCT Number); 2023-510381-28-01 (Registry Identifier: CTIS European Clinical Trial Identification System)
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Surgical Complication
Keywords: tranexamic acid postoperative bleeding infection wound rupture seroma thromboembolism
MeSH Terms: interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized controlled prospective interventional trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identically shaped ampoules containing traneamic acid (Cyklokapron, Pfizer) and 0.9% Saline (Lavoisier, France) have been identified. The ampoule top part is camouflaged with a tight-fitting black tube which preserves the breaking point on the neck of the ampoule. The ampoules will be re-labeled with study-specific labels (text will be in accordance with Regulation 546/2014, annex VI). Randomized study envelopes will be provided in packages of two, with a 1:1 TXA:Placebo randomization, enabling a within-patient randomization in bilateral procedures.
  Randomization, blinding, labelling, shipment of ampoules and keeping of the randomization code will be done by Smerud Medical Research International AS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid arm (Active Comparator): Anonymous ampoule containing 5 ml of 100 mg/ml Tranexamic Acid. If surgeon wants to apply tranexamic acid onto the wound surface, the study ampoule will be diluted and applied in accordance with the surgeon's practice when using Tranexamic Acid.
  Interventions: Drug: Tranexamic Acid 100 MG/ML
- Placebo arm (Placebo Comparator): Anonymous ampoule containing 5 ml of 0.9% NaCl. If surgeon wants to apply tranexamic acid onto the wound surface, the study ampoule will be diluted and applied in accordance with the surgeon's practice when using Tranexamic Acid.
  Interventions: Drug: 0.9%sodium chloride

INTERVENTIONS:
Drug: Tranexamic Acid 100 MG/ML — If surgeon wants to apply tranexamic acid onto the wound surface, the study ampoule will be diluted and applied in accordance with the surgeon's practice when using tranexamic acid
  Other Names: Saline (placebo)
  Arms: Tranexamic acid arm
Drug: 0.9%sodium chloride — If surgeon wants to apply tranexamic acid onto the wound surface, the study ampoule will be diluted and applied in accordance with the surgeon's practice when using Tranexamic Acid.
  Arms: Placebo arm

SUMMARY:
Study objective:

This is a study to investigate whether applying the drug tranexamic acid (TXA) onto a surgical wound surface may affect the incidence of surgical complications such as re-bleeding needing intervention, wound complications such as infection, wound rupture or seroma, or if it may increase the risk of blood clots.

Eligible patients:

Patients undergoing plastic surgical procedures with wounds that would normally receive application of TXA to reduce bleeding after surgery.

Study intervention:

Participants will receive a single local application of study drug onto their wound surfaces at the end of surgery. Study drug will be identical looking ampoules which contain either TXA or placebo (saline). Neither participants nor study personnel will know the contents of the ampoules.

DETAILED DESCRIPTION:
Any serious postoperative complication needing intervention, specifically re-bleeding, wound infection, wound rupture, or the occurrence of blood clots for the first 30 days after surgery will be registered through the following interventions:

* Screening of patient medical records
* Distribution of an electronic self-report form (eForsk®) to participating patients at postoperative day 30
* Follow-up phone call to verify data after day 30.

The study is terminated after the final phone call. All study data will be registered in an electronic, pseudonymous web-based registration form (eCRF/Viedoc®).

Number of participants: To assess the effect of TXA on the defined surgical complications compared to placebo, 1500 patients are needed in each group.

Data monitoring committee:

A data monitoring committee consisting of a group of independent scientists will be appointed for this study to monitor the safety and scientific integrity of this human research intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible to be included in the study only if all of the following criteria apply:

  1. They are to undergo a surgical procedure within the field of plastic surgery where the procedure involves use of topical TXA at the participating center.
  2. They are over 18 years of age and capable of independently providing informed consent
  3. They have received adequate oral and written information about the study and signed the informed-consent form

Exclusion Criteria:

* Patients with known allergy to tranexamic acid. Insufficient knowledge of national language or English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative re-bleeding | 10 days
  • Comparison between wounds receiving TXA versus placebo of the incidence of postoperative re-bleeding within the first postoperative 10 days

SECONDARY OUTCOMES:
Postoperative wound infection | 30 days
  • Comparison between wounds receiving TXA versus placebo of the incidence of postoperative wound infection within the first 30 days requiring any of the following: Extra outpatient follow-up, re-operation, or revision or antibiotic treatment.
Postoperative wound rupture | 30 days
  • Comparison between wounds receiving TXA versus placebo of the incidence of wound rupture within the first 30 days requiring any of the following: Extra outpatient follow-up, re-operation, or revision.
Postoperative thromboembolic events | 30 days
  • Comparison between wounds receiving TXA versus placebo of the incidence of • thromboembolic events defined as thrombophlebitis, deep venous thrombosis, pulmonary embolus, cerebral or coronary infarctions until 30 days postoperatively
Postoperative seroma | Between day 10 and 30
  • Comparison between wounds receiving TXA versus placebo of the incidence of • seroma defined as the need for aspiration of fluids, or spontaneous evacuation of voluminous fluids, between 10 and 30 days postoperatively
Any other postoperative complication | 30 days
  • Comparison between wounds receiving TXA versus placebo of the incidence of • other possible adverse effects causing contact with the health service until 30 days postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Kjersti Ausen, MD PhD, Principal Investigator — St Olav's University Hospital
Locations (1):
- St Olav's University Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data can be made available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available after the completion and publication of the study and will remain available upon reasonable request. Data will be stored for 25 years.
Access Criteria: First or last author must be contacted with a detailed description of what data is needed for. Whether data will be shared must be determined by the investigators and possibly by the regional ethic committee.